CLINICAL TRIAL: NCT01156597
Title: Effects of Pioglitazone on Reverse Cholesterol Transport and HDL Function in Persons With Diabetes
Brief Title: Effects of Pioglitazone on High-density Lipoprotein (HDL) Function in Persons With Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Armando J Mendez, Research Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 06-009A
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; dyslipidemia; pioglitazone; HDL-Cholesterol; Reverse cholesterol transport
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Dyslipidemias | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone Group (Active Comparator): This is a baseline versus treatment study comparing subjects on pioglitazone to a matched group of subjects treated with either metformin or sulfonylurea with the intent of controlling blood sugar to a comparable level
  Interventions: Drug: pioglitazone
- Comparator Group (No Intervention): This group of subjects will be maintained on standard treatment with either metformin or sulfonylurea with the intent of controlling blood sugar to a comparable level as group treated with pioglitazone.

INTERVENTIONS:
Drug: pioglitazone — 30 mg daily for three weeks increase to 45 mg daily for 21 more weeks
  Other Names: ACTOS
  Arms: Pioglitazone Group

SUMMARY:
Metabolic defects contributing to the development of type 2 diabetes (T2D) are relative insulin insufficiency and insulin resistance that are associated with a cluster of abnormalities that increase the risk for cardiovascular disease including dyslipidemia, inflammation, hemodynamic changes and endothelial dysfunction. The dyslipidemia associated with T2D is characterized by elevated triglycerides and decreased high-density lipoprotein-cholesterol (HDL). The ability of the insulin sensitizing agent pioglitazone (ACTOS®) , to improve hyperglycemia in subjects with T2D is now well established. Pioglitazone functions as a PPAR-γ (peroxisome proliferator-activated receptor gamma) agonists and this class of drugs have demonstrated several other potential benefits, beyond glucose homeostasis. Specifically pioglitazone can improve diabetic dyslipidemia by increasing HDL cholesterol and lowing triglycerides. A potential beneficial effect on reverse cholesterol transport may be mediated by the increased HDL levels. This proposal aims to examine the effect of PPAR-γ activation by PIO on various aspects of reverse cholesterol transport by testing the hypothesis that PIO treatment affects key steps in the reverse cholesterol transport pathway either directly, through induction of protein expression, or indirectly, by altering HDL structure and composition leading to increase cholesterol flux through this pathway.

DETAILED DESCRIPTION:
Thiazolidinediones (TZDs) are pharmacological ligands for the nuclear receptor peroxisome-proliferator-activated receptor gamma (PPAR-γ). When activated, the receptor binds with response elements on DNA, altering transcription of a variety of genes that regulate carbohydrate and lipid metabolism1. The hypoglycemic and insulin sensitizing effects of PIO and other TZD compounds are well established2-4. The most prominent effect is increased insulin-stimulated glucose uptake by skeletal muscle cells5,6. The receptor is most highly expressed in adipocytes, while expression in myocytes is comparatively minor. Therefore, the increase in glucose uptake by muscle may largely be an indirect effect mediated through TZD interaction with adipocytes7-9. Candidates for the intermediary signal between fat and muscle include leptin, free fatty acids, tumor necrosis factor-α, adiponectin, and resistin.

T2D is associated with a cluster of lipid and lipoprotein abnormalities including reduced HDL, elevated triglycerides and a predominance of small dense LDL particles10. Altered metabolism of triglyceride rich lipoproteins is crucial in the pathophysiology of diabetic dyslipidemia. Alterations include increased hepatic production and delayed clearance from plasma of large very low density lipoproteins (VLDL) and intestinal chylomicrons. Increased levels of these particles also results in increased production of small dense low density lipoprotein (LDL). The reduction in high density lipoprotein (HDL) associated with T2D appears related to CETP-mediated transfer of cholesterol from HDL to triglyceride rich particles in exchange for triglyceride. The triglyceride rich HDL are hydrolyzed by hepatic lipase, reducing particles size, then more rapidly cleared from the circulation11. Reduced HDL is due to mostly a decrease in HDL2, however, there are increased levels of small HDL3 12.

In addition to their ability to induce insulin sensitivity in T2D subjects, TZDs also have certain lipid benefits. HDL cholesterol concentrations are often increased with TZD therapy and triglyceride concentrations frequently fall13. A nonrandomized clinical comparison of potential differences in lipid effects among TZDs14 demonstrated the beneficial effect on lipids was most with pioglitazone (PIO) and least with rosiglitazone (ROSI)15. These observations were confirmed in a study investigating the lipid-lowering effects of TZDs showing that PIO was associated with significantly greater improvements in triglycerides, HDL cholesterol, non-HDL cholesterol, and LDL particle size compared with ROSI 16. The mechanism(s) by which these agents exert differential effects on the lipid profile are not clearly understood. Whether these differences in lipid effects translate into differences for the risk of CVD is not clear. Trials to determine the effects of pioglitazone and rosiglitazone on CVD outcomes are underway and should identify any cardiovascular benefits of the two drugs.

Lipid metabolism plays a central role in the development of atherosclerosis. Elevated LDL and decreased HDL cholesterol are important risk factors for the development of coronary artery disease (CAD). The major cholesterol-carrying lipoprotein in the blood is LDL and many studies have shown the independent relationship between LDL cholesterol and atherosclerosis in both non-diabetic and diabetic subjects17. The metabolism of HDL, which are inversely related to risk of atherosclerotic cardiovascular disease, involves a complex interplay of factors regulating HDL synthesis, intravascular remodeling, and catabolism18. The anti-atherogenic property of HDL has been attributed, at least in part, to the ability of HDL to promote cholesterol removal (efflux) from cells, the first step in the reverse cholesterol transport pathway 19.

Reduced HDL in T2D results from increased clearance of small HDL particles20, and PIO treatment of these subjects raises HDL levels by 10-15% through as yet poorly defined mechanisms. Studies by Ginsberg and colleagues21, in an elegant study, examined the effects PIO treatment in patients with T2D on various aspects of lipoprotein metabolism. PIO raised HDL cholesterol levels 14%, but no change in apoA-I production rates, or fall in apoA-I synthetic rates were observed during PIO therapy22. ApoA-I synthesis is regulated by several transcription factors, including PPAR-α; there is no evidence that PPAR-α plays a role in apoA-I synthesis in vivo, although both PIO and ROSI have been reported to stimulate apoA-I secretion from HepG2 cells23. The authors suggest that the rise in HDL may have resulted from reduced CETP-mediated exchange of VLDL triglycerides for HDL cholesterol, concomitant with the PIO-associated fall in VLDL levels or a reduced the mass or activity of HL thus increasing HDL levels. There are no published data regarding PPAR-γ agonists on HL activity, but the authors found no change in HL mass in preheparin serum by PIO treatment. A final possibility proposed by these authors was PPAR-γ signaling may play a role in stimulating expression of the gene encoding ABCA1 which could increase the flux of cholesterol from cells onto nascent apoA-I.

Study Aims Characterize the structural and functional changes in plasma lipids and lipoproteins in T2D subjects before and after PIO treatment. A major emphasis will compare serum HDL function as related to reverse cholesterol transport by plasma lipoproteins at baseline and after PIO treatment.

We hypothesize that increased levels of HDL resulting from PIO therapy will affect particle size, density distribution and the lipid and lipoprotein composition of HDL and that such changes may alter the activity of several key steps involved in reverse cholesterol transport, namely the ability to promote cellular cholesterol efflux, cholesterol esterification by LCAT and transport of esterified cholesterol from HDL to the apoB containing lipoproteins.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, men and women, WHO criteria, aged 35-70 years
* HbA1c 7.5-10.0%
* BMI 26-39 Kg/m2
* Either receiving dietary therapy only or monotherapy with either sulfonylurea or metformin
* Already on statin therapy

Exclusion Criteria:

* Cardiovascular disease
* Renal disease
* Other systemic disease
* Abnormal liver function tests (ALT or AST>1.5 X ULN)
* Uncontrolled hypertension (BP >160/110)
* Triglyceride levels >400 mg/dl
* Lipid modifying drugs; fibrates, ezetimibe, niacin, bile sequestrants, but not statins (see below),
* Estrogen treatment or thyroid disease
* Psychiatric condition or substance abuse

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armando J Mendez, PhD, Principal Investigator — University of Miami; Ronald Goldberg, MD, Principal Investigator — University of Miami
Locations (1):
- Diabetes Research Institute, Miami, Florida, United States

REFERENCES:
- [Background] Mudaliar S, Henry RR. New oral therapies for type 2 diabetes mellitus: The glitazones or insulin sensitizers. Annu Rev Med. 2001;52:239-57. doi: 10.1146/annurev.med.52.1.239. PMID 11160777
- [Background] Campbell IW. Long-term glycaemic control with pioglitazone in patients with type 2 diabetes. Int J Clin Pract. 2004 Feb;58(2):192-200. doi: 10.1111/j.1368-5031.2004.0108.x. PMID 15055868
- [Background] Olansky L, Marchetti A, Lau H. Multicenter retrospective assessment of thiazolidinedione monotherapy and combination therapy in patients with type 2 diabetes: comparative subgroup analyses of glycemic control and blood lipid levels. Clin Ther. 2003;25 Suppl B:B64-80. doi: 10.1016/s0149-2918(03)80243-6. PMID 14553867
- [Background] Charbonnel B, Roden M, Urquhart R, Mariz S, Johns D, Mihm M, Widel M, Tan M. Pioglitazone elicits long-term improvements in insulin sensitivity in patients with type 2 diabetes: comparisons with gliclazide-based regimens. Diabetologia. 2005 Mar;48(3):553-60. doi: 10.1007/s00125-004-1651-9. Epub 2005 Mar 1. PMID 15739120
- [Background] Rasouli N, Raue U, Miles LM, Lu T, Di Gregorio GB, Elbein SC, Kern PA. Pioglitazone improves insulin sensitivity through reduction in muscle lipid and redistribution of lipid into adipose tissue. Am J Physiol Endocrinol Metab. 2005 May;288(5):E930-4. doi: 10.1152/ajpendo.00522.2004. Epub 2005 Jan 4. PMID 15632102

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pioglitazone Group | Comparator Group
Started | 16 | 14
Completed | 13 | 13
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pioglitazone Group: This is a baseline versus treatment study comparing subjects on pioglitazone to a matched group of subjects treated with either metformin or sulfonylurea with the intent of controlling blood sugar to a comparable level
  The pioglitazone treatment regimen for this arm of the study: 30 mg daily for three weeks increase to 45 mg daily for 21 more weeks
- Total: Total of all reporting groups
Arm/Group | Pioglitazone Group | Comparator Group | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (5.9) | 58.2 (8.2) | 58.3 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30
Hemoglobin A1C [Mean (Standard Deviation); unit: %] | 7.2 (1.3) | 7.8 (1.3) | 7.5 (1.2)
High Density Lipoprotein [Mean (Standard Deviation); unit: mg/dl] | 45.3 (11.2) | 48.0 (8.4) | 46.7 (9.8)

OUTCOME MEASURES:

1. Primary Outcome: Increased HDL-Cholesterol and Decreased Triglycerides
Description: The primary endpoint will be increased high density lipoprotein cholesterol and decreased triglycerides measured as the difference after 12 or 24 weeks of treatment from baseline levels. The data are expressed as the percent change from the baseline value and calculated using he equation:
  * Change=[100%*(Endpoint value - Baseline Value)/Baseline Value]
Time Frame: 24 weeks
Population: All subjects that completed the study were used for the final analysis
Measure: Mean (Standard Deviation); unit: % Change
Arm/Group | Pioglitazone Group | Comparator Group
Number analyzed (Participants) | 13 | 13
% Change
  % Change in HDL cholesterol at 12 weeks | 7.9 (15.3) | 2.7 (9.9)
  % Change in HDL cholesterol at 24 weeks | 15.7 (5.9) | -1.5 (3.8)
  % Change in triglycerides at 12 weeks | -10.9 (26.6) | 7.4 (33.5)
  % Change in triglycerides at 24 weeks | -15.4 (6.3) | 19.7 (11.3)
Statistical Analysis 1: Comparison: Pioglitazone Group vs Comparator Group; Test type: Superiority or Other; p = 0.05, ANOVA; The percent change of HDL and triglycerides from baseline between groups was evaluated by ANOVA using baseline, 12 week and 24 week values

2. Secondary Outcome: HDL Apolipoprotein Levels at Study End-point
Description: Lipoproteins will be isolated and analyzed using the gradient ultracentrifugation-high pressure liquid chromatography technique to isolate very low-density lipoprotein (VLDL), intermediate density lipoprotein (IDL), LDL, and high density lipoprotein (HDL) subfractions. Protein and lipid compositions of HDL is determined
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone Group | Comparator Group
Number analyzed (Participants) | 13 | 13
mg/dL
  HDL-apoAI at end point | 65.0 (0.9) | 65.7 (7.0)
  HDL-apoAII at end point | 26.6 (4.8) | 22.6 (4.3)
  HDL-apoCI at end point | 10.9 (2.2) | 8.4 (2.5)
  HDL-apoCII at end point | 3.5 (1.3) | 2.8 (1.3)
  HDL-apoCIII at end point | 11.8 (4.0) | 12.5 (2.6)
  HDL-apoM at end point | 0.62 (0.2) | 0.43 (0.2)

3. Secondary Outcome: Cholesterol Efflux Capacity of HDL
Description: The ability of serum HDL to remove cholesterol from cultured cells will be assessed as an in vitro method to evaluate a functional changes in HDL mediated by changes due to pioglitazone treatment. Cells were incubated with 2% serum from each study subject diluted in culture medium and incubations were performed for a total of 4 hours. Cholesterol efflux was calculated as the percent of cholesterol removed from the cells and appearing in the culture medium normalized to a reference serum pool as described in detail by de la Llera-Moya et al (de la Llera-Moya M, Drazul-Schrader D, Asztalos BF, Cuchel M, Rader DJ, Rothblat GH. The ability to promote efflux via ABCA1 determines the capacity of serum specimens with similar high-density lipoprotein cholesterol to remove cholesterol from macrophages. Arterioscler Thromb Vasc Biol. 2010 Apr;30(4):796-801. doi: 10.1161/ATVBAHA.109.199158. PMID: 20075420).
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Pioglitazone Group | Comparator Group
Number analyzed (Participants) | 13 | 13
Ratio | 1.02 (0.10) | 1.05 (0.07)

ADVERSE EVENTS:
Arm/Group | Pioglitazone Group | Comparator Group
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less